CLINICAL TRIAL: NCT01370252
Title: Arthroscopic Ankle Arthrodesis: Measuring Post-operative Pain to Assess the Potential for Outpatient Surgery.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hammond, Allan, M.D. (Individual)
Responsible Party: Dr. Allan Hammond, University of Manitoba, Assistant Professor, Faculty of Medicine
Other Study IDs: H2011:070
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis
Keywords: ankle arthrodesis; pain; arthroscopic technique; ankle osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- scope technique
- open technique

SUMMARY:
Post-operative pain will be measured using a pain diary for one week post-surgery. The purpose is to test the assumption that the arthroscopic technique leads to less post-operative pain and results in shorter hospital stays when compared to the open technique. It is believed that the arthroscopic technique will result in minimal pain when compared to the open technique, allowing this procedure to be performed as day surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ankle osteoarthritis with adequate bone stock

Exclusion Criteria:

* Mental or physical inability to consent or answer pain questions, pre-operative or peri-operative morbidity impairing mobility, pre-operative opioid therapy, non-steroidal anti-inflammatory drugs or steroids within 24 hours before skin incision, kidney or liver dysfunction, morbid obesity, smoking, significant bony deformity, significant loss of bone stock or diabetes with sensory changes will be cause for exclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients selected from the surgeons waitlist.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-06

PRIMARY OUTCOMES:
Numeric Rating Pain Scale (NRPS) | recorded for one week post-operatively
  A scale from 0-10 is used for patients to record the amount of pain they are experiencing at a given time. Multiple questions are asked on a daily basis in a pain diary to report pain in the morning, at night, with movement, before and after pain medication.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Hammond, MD, FRCSC, Principal Investigator — University of Manitoba, Faculty of Medicine, Department of Orthopedics, Assistant professor
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada